CLINICAL TRIAL: NCT06866509
Title: A Prospective, Multicenter, Non-Interventional Observational Study to Investigate Changes in Blood Lipid Levels and Safety Following Administration of Litorvazet® Tablets in Patients With Dyslipidemia
Brief Title: To Investigate Blood Lipid Changes and Safety After Litorvazet® Tablets in Dyslipidemia Patients
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWLTV_OS_01
Record Dates: First submitted 2025-01-20; First posted 2025-03-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Dyslipidemia: Patients With Dyslipidemia
  Interventions: Drug: Litorvazet Tablet 10/10mg; Drug: Litorvazet Tablet10/20mg; Drug: Litorvazet Tablet 10/40mg

INTERVENTIONS:
Drug: Litorvazet Tablet 10/10mg — Ezetimibe 10 mg + Atorvastatin 10 mg
Drug: Litorvazet Tablet10/20mg — Ezetimibe 10 mg + Atorvastatin 20 mg
Drug: Litorvazet Tablet 10/40mg — Ezetimibe 10 mg + Atorvastatin 40 mg

SUMMARY:
This study aims to investigate the lipid-lowering effects and safety of administering Litorvazet tablets (ezetimibe/atorvastatin) over a 24-week period in patients with dyslipidemia scheduled to receive Litorvazet tablets in a real-world clinical setting.

DETAILED DESCRIPTION:
In a real-world clinical setting, Litorvazet® tablets will be administered to patients based on the investigator's medical judgment in accordance with the approved prescribing information (indications, dosage, and administration, precautions for use, etc.).

Participants for data collection in this study will be patients diagnosed with dyslipidemia as determined by the judgment of their attending physician.

All treatments, including drug administration and clinical laboratory tests conducted after the administration of Litorvazet® tablets, will be carried out based solely on the investigator's (attending physician's) medical judgment and will not be influenced by the patient's participation in the study. Information relevant to this observational study will be collected for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 19 years or older at the time of the screening visit.
* Patients with dyslipidemia who are scheduled to receive Litorvazet® tablets based on the investigator's (treating physician's) medical judgment and in accordance with the approved indications.
* Individuals who have voluntarily provided written consent to participate in this study.

Exclusion Criteria:

* Individuals who meet any contraindications for Litorvazet® tablets as specified in the product labeling:
* Those with hypersensitivity to any components of this medication.
* Patients with active liver disease or those with persistently elevated serum transaminase levels of unknown cause.
* Patients with muscle disorders.
* Pregnant women, women who may be pregnant, or breastfeeding mothers.
* Women of childbearing potential who are not using appropriate contraceptive methods.
* Patients receiving glecaprevir and pibrentasvir.
* Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Individuals with a history of receiving Litorvazett® tablets prior to participating in this study.
* Individuals deemed unsuitable for participation in this observational study by the investigator (treating physician) for reasons beyond those listed above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To estimate LDL-C changes at Week 24 in a dyslipidemia population on Ezetimibe/Atorvastatin, clinical trial data from participants with similar baseline conditions were used. The standard deviation (SD) of LDL-C changes ranged from 23.57 to 38.91 mg/dL in two studies, and a pooled SD was calculated.
  With a 20% dropout rate, 3,000 participants (2,400 evaluable) were included. Assuming an SD of 33 mg/dL for LDL-C changes, a two-sided 95% confidence interval with a 1.32 mg/dL margin of error was generated. Including the dropout rate, a total of 3,000 participants were selected.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in LDL-C Levels Compared to Baseline | at Week 24
  Change in LDL-C Levels at Week 24 Compared to Baseline

SECONDARY OUTCOMES:
Changes in LDL-C levels compared to baseline [excluding primary endpoints]. | at Week 12
  Changes in LDL-C levels at Week 12 compared to baseline [excluding primary endpoints].
Percentage changes (%) in LDL-C levels compared to baseline [excluding primary endpoints]. | at Week 12
  Percentage changes (%) in LDL-C levels at Week 12 compared to baseline [excluding primary endpoints].
Changes in LDL-C levels compared to baseline [excluding primary endpoints]. | at Week 24
  Changes in LDL-C levels at Week 24 compared to baseline [excluding primary endpoints].
Percentage changes (%) in LDL-C levels compared to baseline [excluding primary endpoints]. | at Week 24
  Percentage changes (%) in LDL-C levels at Week 24 compared to baseline [excluding primary endpoints].
Changes in HDL-C levels compared to baseline | at Week 12
  Changes in HDL-C levels at Week 12 compared to baseline.
Percentage changes (%) in HDL-C levels compared to baseline | at Week 12
  Percentage changes (%) in HDL-C levels at Week 12 compared to baseline.
Changes in HDL-C levels compared to baseline | at Week 24
  Changes in HDL-C levels at Week 24 compared to baseline.
Percentage changes (%) in HDL-C levels compared to baseline | at Week 24
  Percentage changes (%) in HDL-C levels at Week 24 compared to baseline.
Changes in Non-HDL-C levels compared to baseline | at Week 12
  Changes in Non-HDL-C levels at Week 12 compared to baseline
Percentage changes (%) in Non-HDL-C levels compared to baseline | at Week 12
  Percentage changes (%) in Non-HDL-C levels at Week 12 compared to baseline
Changes in Non-HDL-C levels compared to baseline | at Week 24
  Changes in Non-HDL-C levels at Week 24 compared to baseline
Percentage changes (%) in Non-HDL-C levels compared to baseline | at Week 24
  Percentage changes (%) in Non-HDL-C levels at Week 24 compared to baseline
Changes in TG levels compared to baseline | at Week 12
  Changes in TG levels at Week 12 compared to baseline.
Percentage changes (%) in TG levels compared to baseline | at Week 12
  Percentage changes (%) in TG levels at Week 12 compared to baseline.
Changes in TG levels compared to baseline | at Week 24
  Changes in TG levels at Week 24 compared to baseline
Percentage changes (%) in TG levels compared to baseline | at Week 24
  Percentage changes (%) in TG levels at Week 24 compared to baseline
Changes in TC levels compared to baseline | at Week 12
  Changes in TC levels at Week 12 compared to baseline
Percentage changes (%) in TC levels compared to baseline | at Week 12
  Percentage changes (%) in TC levels at Week 12 compared to baseline
Changes in TC levels compared to baseline | at Week 24
  Changes in TC levels at Week 24 compared to baseline
Percentage changes (%) in TC levels compared to baseline | at Week 24
  Percentage changes (%) in TC levels at Week 24 compared to baseline
Changes in ALT levels compared to baseline | at Week 12
  Changes in ALT levels at Week 12 compared to baseline
Changes in AST levels compared to baseline | at Week 12
  Changes in AST levels at Week 12 compared to baseline
Percentage changes (%) in ALT levels compared to baseline | at Week 12
  Percentage changes (%) in ALT levels at Week 12 compared to baseline
Percentage changes (%) in AST levels compared to baseline | at Week 12
  Percentage changes (%) in AST levels at Week 12 compared to baseline
Changes in ALT levels compared to baseline | at Week 24
  Changes in ALT levels at Week 24 compared to baseline
Changes in AST levels compared to baseline | at Week 24
  Changes in AST levels at Week 24 compared to baseline
Percentage changes (%) in ALT levels compared to baseline | at Week 24
  Percentage changes (%) in ALT levels at Week 24 compared to baseline
Percentage changes (%) in AST levels compared to baseline | at Week 24
  Percentage changes (%) in AST levels at Week 24 compared to baseline
Changes in systolic blood pressure compared to baseline | at Week 12
  Changes in systolic blood pressure at Week 12 compared to baseline
Changes in diastolic blood pressure compared to baseline | at Week 12
  Changes in diastolic blood pressure at Week 12 compared to baseline
Percentage changes (%) in systolic blood pressure compared to baseline | at Week 12
  Percentage changes (%) in systolic blood pressure at Week 12 compared to baseline
Percentage changes (%) in diastolic blood pressure compared to baseline | at Week 12
  Percentage changes (%) in diastolic blood pressure at Week 12 compared to baseline
Changes in systolic blood pressure compared to baseline | at Week 24
  Changes in systolic blood pressure at Week 24 compared to baseline
Changes in diastolic blood pressure compared to baseline | at Week 24
  Changes in diastolic blood pressure at Week 24 compared to baseline
Percentage changes (%) in systolic blood pressure compared to baseline | at Week 24
  Percentage changes (%) in systolic blood pressure at Week 24 compared to baseline
Percentage changes (%) in diastolic blood pressure compared to baseline | at Week 24
  Percentage changes (%) in diastolic blood pressure at Week 24 compared to baseline
Changes in HbA1c levels compared to baseline | at Week 12
  Changes in HbA1c levels at Week 12 compared to baseline
Percentage changes (%) in HbA1c levels compared to baseline | at Week 12
  Percentage changes (%) in HbA1c levels at Week 12 compared to baseline
Changes in HbA1c levels compared to baseline | at Week 24
  Changes in HbA1c levels at Week 24 compared to baseline
Percentage changes (%) in HbA1c levels compared to baseline | at Week 24
  Percentage changes (%) in HbA1c levels at Week 24 compared to baseline
Changes in LDL-C levels in patients who did not achieve their therapeutic targets based on baseline risk levels | at Week 12
  Changes in LDL-C levels at Week 12 in patients who did not achieve their therapeutic targets based on baseline risk levels
Goal attainment rates in patients who did not achieve their therapeutic targets based on baseline risk levels | at Week 12
  Goal attainment rates at Week 12 in patients who did not achieve their therapeutic targets based on baseline risk levels
Changes in LDL-C levels in patients who did not achieve their therapeutic targets based on baseline risk levels | at Week 24
  Changes in LDL-C levels at Week 24 in patients who did not achieve their therapeutic targets based on baseline risk levels
Goal attainment rates in patients who did not achieve their therapeutic targets based on baseline risk levels | at Week 24
  Goal attainment rates at Week 24 in patients who did not achieve their therapeutic targets based on baseline risk levels
Changes in LDL-C levels in patients who achieved their therapeutic targets based on baseline risk levels | at Week 12
  Changes in LDL-C levels at Week 12 in patients who achieved their therapeutic targets based on baseline risk levels
Goal maintenance rates in patients who achieved their therapeutic targets based on baseline risk levels | at Week 12
  Goal maintenance rates at Week 12 in patients who achieved their therapeutic targets based on baseline risk levels
Changes in LDL-C levels in patients who achieved their therapeutic targets based on baseline risk levels | at Week 24
  Changes in LDL-C levels at Week 24 in patients who achieved their therapeutic targets based on baseline risk levels
Goal maintenance rates in patients who achieved their therapeutic targets based on baseline risk levels | at Week 24
  Goal maintenance rates at Week 24 in patients who achieved their therapeutic targets based on baseline risk levels
Changes in LDL-C levels in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 12
  Changes in LDL-C levels at Week 12 in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Goal maintenance rates in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 12
  Goal maintenance rates at Week 12 in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Changes in LDL-C levels in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 24
  Changes in LDL-C levels at Week 24 in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Goal maintenance rates in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 24
  Goal maintenance rates at Week 24 in patients who achieved their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Changes in LDL-C levels in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 12
  Changes in LDL-C levels at Week 12 in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Goal attainment rates in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 12
  Goal attainment rates at Week 12 in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Changes in LDL-C levels in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 24
  Changes in LDL-C levels at Week 24 in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment
Goal attainment rates in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment | at Week 24
  Goal attainment rates at Week 24 in patients who did not achieve their therapeutic targets based on baseline risk levels, categorized by the previously administered dyslipidemia treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Mi Park, Dr., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea